CLINICAL TRIAL: NCT06605937
Title: Eustachian Dysfunction Occurring After Adenoidectomy and/or Adenotonsillectomy and the Effect of Postoperative Eustachian Milking Maneuver on Eustachian Dysfunction
Brief Title: The Effect of Postoperative Eustachian Milking Maneuver on Eustachian Tube Dysfunction
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 04-2024/03
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Middle Ear Pressure; Otalgia
Keywords: Eustachian Milking Maneuver; Analgesia; Eustachian dysfunction
MeSH Terms: conditions — Earache; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Grup 1: The children undergoing adenoidectomy and/or adenotonsillectomy whose parents will apply eustachian milking maneuver in the post-operative period.
  Interventions: Other: Eustachian milking maneuver with routine postoperative treatment protocol; Other: Routine postoperative treatment protocol
- Grup 2: The children undergoing adenoidectomy and/or adenotonsillectomy whose parents will not apply eustachian milking maneuvers in the post-operative period.
  Interventions: Other: Routine postoperative treatment protocol

INTERVENTIONS:
Other: Eustachian milking maneuver with routine postoperative treatment protocol — Eustachian milking maneuver will be applied by the patients parents 3 times a day for 7 days in the post-operative period.
  Groups: Grup 1
Other: Routine postoperative treatment protocol — The children adenoidectomy and/or adenotonsillectomy whose parents will not apply eustachian healing maneuvers in the post-operative period.

SUMMARY:
This study will evaluate the effectiveness of this lymphatic drainage method in eliminating otalgia interruption due to eustachian dysfunction and reducing middle ear pressure, which occurs in the postoperative period after adenoidectomy and/or adenotonsillectomy.

DETAILED DESCRIPTION:
The eustachian tube lies between the middle ear and the nasopharyngeal cavity and provides ventilation of the middle ear. The most important function of the Eustachian tube is to balance the air pressure in the middle ear with atmospheric pressure.

Temporary eustachian dysfunction and ear fullness occur in the early postoperative period after adenoidectomy and/or adenotonsillectomy. This temporary eustachian dysfunction is considered to be caused by clots and edema in the nasopharynx after surgery. In addition, trauma to the eustachian tube during adenoidectomy performed by curettage also contributes.

Eustachian dysfunction may present at the post-operative period resulted in otalgia related to middle ear pressure in the pediatric patients undergoing adenoidectomy or adenotonsillectomy. In this case, the need for analgesic agents rises in the early postoperative operiod and beyond this stituation impairs the quality of the healing process.

Reducing middle ear pressure by ensuring the mobility of the eustachian tube with the eustachian milking maneuver, which is a lymphatic drainage method, may reduce the otalgia symptoms during the post-operative recovery period, thus reducing the use of analgesic agents and improving the quality of the healing process. The aim of this observational study is to investigate to what extent a eustachian therapy maneuver corrects the negative values in middle ear pressure in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

Patients with ASA 1 and 2 The parent will be able to perform eustachian milking manoeuvres

Exclusion Criteria:

Tympanometric examination performed in the preoperative period revealed eustachian dysfunction Craniofacial malformation

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 80 patients aged 3-15 years who were indicated for adenoidectomy and/or adenotonsillectomy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Middle ear pressure | Perioperative period
  Tympanometry is an objective test of middle-ear function. The test is performed by inserting the tympanometer probe in the ear canal. The instrument changes the pressure in the ear, generates a pure tone, and measures the eardrum responses to the sound at different pressures. This produces a series of data measuring how admittance varies with pressure, which is plotted as a tympanogram

SECONDARY OUTCOMES:
Evaluation of postoperative otalgia symptoms | Postoperative period
  Postoperative pain related to ear will be evaluated with Visual Analog Scale (VAS). Children will be asked to choose the pain they feel according to the facial expression in the picture. 0 indicates no pain, 10 indicates severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Duran, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Karaman, Turkey (Türkiye)